CLINICAL TRIAL: NCT04039971
Title: Quadriceps Tendon Autograft, Tendon-Bone Versus All-Soft-Tissue for Anterior Cruciate Ligament Reconstruction: A Patient-Blinded Randomized Clinical Trial
Brief Title: Tendon-Bone Versus All-Soft-Tissue for ACL Reconstruction: A Patient-Blinded Randomized Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-1445
Record Dates: First submitted 2019-07-26; First posted 2019-07-31 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear
Keywords: ACL; ACL Tear; ACL Injury; ACL Rupture; Anterior Cruciate Ligament Tear; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament; ACL Repair; ACL Reconstruction; ACL Surgery; Anterior Cruciate Ligament Repair; Anterior Cruciate Ligament Reconstruction; Anterior Cruciate Ligament Surgery
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tendon-Bone Graft (Active Comparator): Participants receive the Quadriceps Tendon Tendon-Bone Graft technique during ACL reconstruction.
  Interventions: Procedure: ACL Reconstruction
- All-Soft-Tissue Graft (Active Comparator): Participants receive the Quadriceps Tendon All-Soft-Tissue Graft technique during ACL reconstruction.
  Interventions: Procedure: ACL Reconstruction

INTERVENTIONS:
Procedure: ACL Reconstruction — Surgical techniques

SUMMARY:
In primary pediatric Anterior cruciate ligament (ACL) reconstruction, the quadriceps tendon with either tendon and patellar bone or an all-tendon graft is commonly employed. However, no randomized control trial has sought to discern the superior graft option in regards to both short-term and long-term patient outcomes.The purpose of this study is to assess the differences between these two widely used surgical techniques in ACL reconstruction by examining short, intermediate, and long term outcomes of both approaches.

DETAILED DESCRIPTION:
It is well known that ACL injuries are among the most common sports and knee injuries. As a result, ACL reconstruction is at the forefront both in terms of research and development and advancements in technique. One focus of research is graft choice and the risks and benefits associated with each. There are multiple valid graft choices including bone-patellar tendon-bone, hamstring tendon, quadriceps tendon, quadriceps tendon-patellar bone, and allograft. Graft choice is often patient centered and based on both patient and surgeon considerations such as age, sex, activity level, surgeon preference and graft associated complications.

The present study seeks to compare the intraoperative, immediate perioperative, intermediate and long-term outcomes between tendon-bone and all-soft-tissue quadriceps tendon autograft in ACL reconstruction in adolescent patients. The investigators will analyze data on operative time, cost, complications, recovery of strength and range of motion, return to sports rates, patient reported outcomes, and failure rates. With this proposal the investigators hope to determine if there is a superior graft technique in this population. Both graft types are validated in the literature separately as options for ACL reconstruction in this age group. There has been no clinical research comparing the two graft types, and therefore no consensus is made among surgeons on whether to use tendon-bone or all-soft-tissue when it comes to the QT autograft. A secondary aim of this study is to obtain patient reported outcomes throughout the post-operative period to determine if the patient experience is different between the two graft types. This data may be used in guiding a surgeon's decision on which type to use with their patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Patients ages 12 to 19 (inclusive)
* Patients undergoing primary ACL reconstruction

Exclusion Criteria:

* Patients with an underlying neuromuscular diagnosis or neurological injury
* Patients with lower extremity fractures, dislocations, or multi-ligamentous injuries, which required surgery, concurrent with or occurring two years or less prior to primary ACL injury.
* Patients with an underlying systemic or musculoskeletal diagnosis

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Short-Term Graft Superiority | 1 to 2 years
  Graft superiority will be evaluated by the time to return to sports and the length of return to sports.
Long-Term Graft Superiority | 5 years
  Long-term graft superiority will be evaluated by graft failure rate or ACL re-rupture.

SECONDARY OUTCOMES:
Patient Reported Outcomes | Pre-operative appointment, 3 months, 6 months, 12 months, 24 months, and 5 years post-operative appointments
  Patients will complete a survey at specific time points to gauge knee function throughout treatment.
Time to Return to Sports Rates | As recorded in post-operative physical therapy visits (approx. 6 months to 1 year)
  Time to return to sports will be evaluated based on physical therapy milestones related to return to sports clearance.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Mayer, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with individuals or organizations outside of the research team.

REFERENCES:
- [Background] Kaeding CC, Pedroza AD, Reinke EK, Huston LJ, Hewett TE, Flanigan DC; MOON Knee Group; Spindler KP. Change in Anterior Cruciate Ligament Graft Choice and Outcomes Over Time. Arthroscopy. 2017 Nov;33(11):2007-2014. doi: 10.1016/j.arthro.2017.06.019. Epub 2017 Aug 26. PMID 28847572
- [Background] Fineberg MS, Zarins B, Sherman OH. Practical considerations in anterior cruciate ligament replacement surgery. Arthroscopy. 2000 Oct;16(7):715-24. doi: 10.1053/jars.2000.8951. PMID 11027755
- [Background] Middleton KK, Hamilton T, Irrgang JJ, Karlsson J, Harner CD, Fu FH. Anatomic anterior cruciate ligament (ACL) reconstruction: a global perspective. Part 1. Knee Surg Sports Traumatol Arthrosc. 2014 Jul;22(7):1467-82. doi: 10.1007/s00167-014-2846-3. Epub 2014 Feb 5. PMID 24497054
- [Background] DeAngelis JP, Fulkerson JP. Quadriceps tendon--a reliable alternative for reconstruction of the anterior cruciate ligament. Clin Sports Med. 2007 Oct;26(4):587-96. doi: 10.1016/j.csm.2007.06.005. PMID 17920954
- [Background] Crall TS, Gilmer BB. Anatomic All-Inside Anterior Cruciate Ligament Reconstruction Using Quadriceps Tendon Autograft. Arthrosc Tech. 2015 Dec 23;4(6):e841-5. doi: 10.1016/j.eats.2015.08.004. eCollection 2015 Dec. PMID 27284521
- [Background] Lee S, Seong SC, Jo CH, Han HS, An JH, Lee MC. Anterior cruciate ligament reconstruction with use of autologous quadriceps tendon graft. J Bone Joint Surg Am. 2007 Oct;89 Suppl 3:116-26. doi: 10.2106/JBJS.G.00632. No abstract available. PMID 17908877
- [Background] Ferrer GA, Miller RM, Murawski CD, Tashman S, Irrgang JJ, Musahl V, Fu FH, Debski RE. Quantitative analysis of the patella following the harvest of a quadriceps tendon autograft with a bone block. Knee Surg Sports Traumatol Arthrosc. 2016 Sep;24(9):2899-2905. doi: 10.1007/s00167-015-3550-7. Epub 2015 Mar 7. PMID 25749653
- [Background] Fink C, Herbort M, Abermann E, Hoser C. Minimally invasive harvest of a quadriceps tendon graft with or without a bone block. Arthrosc Tech. 2014 Aug 11;3(4):e509-13. doi: 10.1016/j.eats.2014.06.003. eCollection 2014 Aug. PMID 25264512
- [Background] Sprowls GR, Robin BN. The Quad Link Technique for an All-Soft-Tissue Quadriceps Graft in Minimally Invasive, All-Inside Anterior Cruciate Ligament Reconstruction. Arthrosc Tech. 2018 Jul 16;7(8):e845-e852. doi: 10.1016/j.eats.2018.04.004. eCollection 2018 Aug. PMID 30167363
- [Background] Schulz AP, Lange V, Gille J, Voigt C, Frohlich S, Stuhr M, Jurgens C. Anterior cruciate ligament reconstruction using bone plug-free quadriceps tendon autograft: intermediate-term clinical outcome after 24-36 months. Open Access J Sports Med. 2013 Nov 19;4:243-9. doi: 10.2147/OAJSM.S49223. eCollection 2013. PMID 24379730
- [Background] Gorschewsky O, Klakow A, Putz A, Mahn H, Neumann W. Clinical comparison of the autologous quadriceps tendon (BQT) and the autologous patella tendon (BPTB) for the reconstruction of the anterior cruciate ligament. Knee Surg Sports Traumatol Arthrosc. 2007 Nov;15(11):1284-92. doi: 10.1007/s00167-007-0371-3. Epub 2007 Aug 25. PMID 17721778
- [Background] Han HS, Seong SC, Lee S, Lee MC. Anterior cruciate ligament reconstruction : quadriceps versus patellar autograft. Clin Orthop Relat Res. 2008 Jan;466(1):198-204. doi: 10.1007/s11999-007-0015-4. Epub 2008 Jan 3. PMID 18196393
- [Background] Kim SJ, Lee SK, Choi CH, Kim SH, Kim SH, Jung M. Graft selection in anterior cruciate ligament reconstruction for smoking patients. Am J Sports Med. 2014 Jan;42(1):166-72. doi: 10.1177/0363546513505191. Epub 2013 Oct 10. PMID 24114749
- [Background] Kim SJ, Kumar P, Oh KS. Anterior cruciate ligament reconstruction: autogenous quadriceps tendon-bone compared with bone-patellar tendon-bone grafts at 2-year follow-up. Arthroscopy. 2009 Feb;25(2):137-44. doi: 10.1016/j.arthro.2008.09.014. Epub 2008 Nov 20. PMID 19171272
- [Background] Streich NA, Barie A, Gotterbarm T, Keil M, Schmitt H. Transphyseal reconstruction of the anterior cruciate ligament in prepubescent athletes. Knee Surg Sports Traumatol Arthrosc. 2010 Nov;18(11):1481-6. doi: 10.1007/s00167-010-1057-9. Epub 2010 Feb 4. PMID 20130837